CLINICAL TRIAL: NCT07332117
Title: A Pilot Study to Assess Body Mass Composition Measurement Using BIA and Muscle Ultrasound in IPF and PPF Patients on Anti-fibrotic Medications
Acronym: AF-BMC
Status: Recruiting | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS ID: 358410
Record Dates: First submitted 2025-09-23; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF); Progressive Pulmonary Fibrosis
Keywords: bioimpedance analysis; muscle ultrasound; body composition
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients to be commenced on anti-fibrotics: Patients with either idiopathic pulmonary fibrosis or progressive pulmonary fibrosis planned to commenced anti-fibrotic medication (either pirfenidone or nintedanib) will be recruited.
  Interventions: Other: No Interventions; Other: No intervention
- Control group: We will also recruit 20 controls with predominantly fibrotic lung disease. Only those with extent of disease > 20% on HRCT as determined by PI and CI will be included. These are patients who in the opinion of the treating physician may require anti-fibrotic treatment in the future, but are not planned to start anti-fibrotic medications over the subsequent 4 months and have not previously been on anti-fibrotic medications.
  Interventions: Other: No Interventions; Other: No intervention

INTERVENTIONS:
Other: No Interventions — No intervention
Other: No intervention — No intervention

SUMMARY:
To assess the impact on body mass composition from anti-fibrotic medications used in fibrotic lung disease by using BIA and muscle ultrasound

DETAILED DESCRIPTION:
This study will be looking at the measurement of body mass composition using bioimpedance analysis (BIA) and quadriceps muscle ultrasound in patients with fibrotic lung disease who are on anti-fibrotic drugs. These anti-fibrotic drugs (nintedanib and pirfenidone) commonly cause gastrointestinal side effects such nausea, loss of appetite and diarrhoea. As a result of these side effects some patients may have a change in the amount of body fat and muscle. This change is not able to be identified using weight or body mass index (BMI). BIA machines are a quick and easy method of looking at body mass composition and require patients to have electrodes attached to their body for approximately 6 seconds. BIA machines are already in routine care for patients with other types of lung conditions. Using muscle ultrasound we will be able to measure the size of the muscle in the thigh.

In addition to the use and tolerability of BIA and muscle ultrasound in this group of patients we will be also taking other measurements including mid-arm circumference and physical tests (sitting to standing, walking speed and muscle strength). We will also use questionnaires to ask about symptoms relating to quality of life, physical activity and gastrointestinal symptoms. Patients will also provide a 3-day diet diary. We will be performing all of the above tests at the beginning before patients start the anti-fibrotic drugs and then again 4 months after starting the drugs and assessing for any changes over this period of time.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Idiopathic pulmonary fibrosis or progressive pulmonary fibrosis
* Newly commencing anti-fibrotic medication (either nintedanib or pirfenidone)
* Subject aged > 18 years
* Able to willingly give consent

Exclusion Criteria:

* Co-morbidities currently requiring enteral feeding
* Weight loss > 10% in preceding 3-6 months
* Significant musculoskeletal issues that may impact muscle mass
* End of life care (expected < 6 weeks left to live)
* Previous anti-fibrotic use
* Currently on > Prednisolone 10mg daily
* Presence of implantable cardioverter defibrillator (ICD) or permanent pacemaker (PPM)
* Heart failure
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being newly commenced on anti-fibrotic medication as part of their clinical care (either nintedanib or pirfenidone)
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Recruitment of patients to study | For study recruitment window of 6 months
  Measured by number of patients consenting/number of patients contacted and rationale for declining
Implementation of study protocol | For the 6 month recruitment window
  Number of patients attending both visits (baseline and 4 months) and rationale for dropout
Feasibility of collection of data | For the the study recruitment window of 6 months
  Collection of data from BIA (skeletal muscle index (SMI), phase angle (PhA) and fat free mass index (FFMI)) and muscle ultrasound (Anterior-posterior diameter of rectus femoris and cross sectional area of rectus femoris)
Acceptability of use of BIA and muscle ultrasound | To be performed at baseline visit and 4 month visit
  Likert scale on use of BIA and muscle ultrasound

SECONDARY OUTCOMES:
Bioelectrical impedance analysis (BIA) | Performed at baseline visit and at 4 month visit
  Messurements taken with BIA include fat-free mass index (FFMI) kg/m2, phase angle (PhA) and skeletal muscle mass (SMM)
Five times sit to stand (5TST) | To be performed at baseline visit and at 4 month visit
  Time taken from moving from sitting to standing position for 5 repetitions will be recorded (seconds)
Four metre gait speed (4MGS) | To be performed at baseline visit and 4 month visit
  Time taken to complete a 4 metre distance walking will be recorded and repeated 3 times (seconds)
Questionnaires assessing gastrointestinal symptoms | To be performed at baseline visit and at 4 month visit
  1. Gastrointestinal symptom rating scale (GSRS) to quantify the severity and impact of gastrointestinal symptoms
  2. Visual analogue scale (VAS) for loss of appetite, nausea and diarrhoea
  3. Past 1 week, how many bowel movements per day
Questionnaires assessing respiratory symptoms and quality of life | To be performed at baseline visit and at 4 month visit
  1) The King's brief interstitial lung disease questionnaire (K-BILD) - a widely validated ILD-specific quality of life questionnaire
Questionnaire to assess levels of physical activity | To be performed at baseline visit and at 4 month visit
  1) International physical activity questionnaire (IPAQ)
Muscle strength | Performed at baseline visit and 4 month visit
  Isometric quadriceps testing - patient seated on a treatment table with hips flexed approximately 85 degrees, thigh is secured to treatment table with one velcro strap placed across thighs, strap attached to patient's ankle and instructed to push their leg forward. This is repeated 3 times with the best reading recorded in kilograms (kg)
Height | To be performed at baseline
  Height - will be taken from the most recent lung function test (within the previous 12 months) in metres (m)
Body weight | Performed at baseline visit and 4 month visit
  Body weight - measured with low clothes and without shoes in kilograms (kg)
Quadriceps ultrasound | To be performed at baseline visit and 4 month visit
  Using phillips (Lumify) linear transducer (C12-4) measurements will be taken by placing the probe perpendicular to the long axis of the the thigh three-fifths of thr distance from the anterior superior iliac spine to the superior patellar border. The average of 3 measurements will be taken of both the anterior-posterior (AP) (cm) and the cross-sectional area of rectus femoris (RFcsa) (cm2). Due to limitations with available software, images will be sent to ImageJ software to determine RFcsa.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Identifiable individual participant data will not be shared with other researchers, however de-identified study results will be submitted to journals for publication.